CLINICAL TRIAL: NCT01497431
Title: Phase I Multiple Dose Study of 12-Week Treatment by Se-Methyl-L-Cysteine(MSC) and L SeMet in Adult Males
Brief Title: Se-Methyl-Seleno-L-Cysteine or Selenomethionine in Preventing Prostate Cancer in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2012-00085; NCI-2012-00085 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000717828; I 182210 (Other: Northwestern University); NWU09-4-03 (Other: DCP); P30CA060553 (NIH); N01CN35157 (NIH)
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: No Evidence of Disease; Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Selenium; selenomethylselenocysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (Se-methyl-seleno L-cysteine) (Experimental): Participants receive Se-methyl-seleno L-cysteine on days 1-84.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Methylselenocysteine
- Arm II (selenomethionine) (Experimental): Participants receive selenomethionine PO on days 1-84.
  Interventions: Dietary Supplement: Selenium; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Arm III (placebo) (Placebo Comparator): Participants receive placebo PO on days 1-84.
  Interventions: Other: Placebo; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Dietary Supplement: Selenium — Given PO
  Other Names: Se
  Arms: Arm II (selenomethionine)
Other: Placebo — Given PO
  Other Names: PLCB
  Arms: Arm III (placebo)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
  Other Names: pharmacological studies
Drug: Methylselenocysteine — Given PO
  Other Names: L-Se-Methylselenocysteine; Methylselenocycteine; MSC; Se-Methyl-seleno-L-cysteine; SeMSC
  Arms: Arm I (Se-methyl-seleno L-cysteine)

SUMMARY:
This randomized phase I trial studies the side effects and the best dose of Se-methyl-seleno-L-cysteine or selenomethionine in preventing prostate cancer in healthy participants. Chemoprevention is the use of certain drugs to keep cancer from forming. The use of Se-methyl-seleno-L-cysteine or selenomethionine, two different types of selenium compounds, may prevent prostate cancer from forming.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the individual toxicity profiles of Se-methyl-seleno-L-cysteine (methyl selenocysteine; MSC) and selenomethionine (SeMet) administered to cohorts of men daily for twelve weeks, with dose escalation with each successive cohort.

SECONDARY OBJECTIVES:

I. To measure the pharmacokinetics of selenium, according to form (MSC vs SeMet): MSC and SeMet impacts on plasma, albumin, and urinary concentrations of selenium over 48 hours on dosing days 1 and 84.

II. To evaluate the pharmacodynamics of selenium by form (MSC vs SeMet): plasma, albumin, and urinary Selenoprotein P (Sepp1) concentrations and glutathione peroxidase (GPx) activity over 48 hours on dosing days 1 and 84.

III. To store plasma and formed elements (red cells plus platelets) for future analysis of methyl selenol and other key selenium species, when those assays become available.

OUTLINE: This is a dose-escalation study. Participants are randomized to 1 of 3 treatment arms.

ARM I: Participants receive Se-methyl-seleno-L-cysteine orally (PO) on days 1-84.

ARM II: Participants receive selenomethionine PO on days 1-84.

ARM III: Participants receive placebo PO on days 1-84.

After completion of study treatment, patients are followed up on day 112.

ELIGIBILITY:
Inclusion Criteria:

* Total body weight between 50 and 115 kg (110 and 250 lbs)
* Hemoglobin (Hgb) > 12 mg/dL
* Platelet count > 100,000/μL
* Absolute neutrophil count (ANC) > 1000/μL
* Creatinine =< institutional upper limit of normal (ULN)
* Serum glutamate pyruvate transaminase (SGPT) and serum glutamic oxaloacetic transaminase (SGOT) < 2.0 x ULN
* Total bilirubin =< ULN (participants with a higher level of bilirubin presumed due to familial metabolism will be considered on an individual basis)
* Life expectancy greater than 3 years
* Participants must agree to use adequate contraception (barrier method of birth control; abstinence) from time of screening until study completion (i.e., for at least 2 weeks after last dose of study drug)
* Ability to understand and the willingness to sign a written informed consent document
* Agree to refrain from use of selenium (Se) supplements (other than the 100 mcg dose common in multivitamins) or Se-containing drugs while on study between 30 days before study drug initiation and Day 84

Exclusion Criteria:

* Not willing to remain at Roswell Park Cancer Institute (RPCI), and in follow up, as required
* Presence of medical conditions which, in the opinion of the investigator, would place either the participant or the integrity of the data at risk
* Serum creatinine > ULN, SGOT or SGPT >= 2.0 x ULN, or bilirubin > ULN
* Treatment with an investigational drug within 30 days prior to the dose of study drug
* Use of selenium [Se] supplements greater than the 100 mcg dose common in multivitamins between 30 days before study drug initiation and Day 84
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to investigational agent (e.g., reaction to other Se supplements)
* Participants who have donated 1 unit of blood within 30 days prior to the first dose of investigational agent
* Eastern Cooperative Oncology Group (ECOG) performance status > 1
* Diagnosed with cancer, other than non-melanoma skin cancer, in last 2 years
* Under treatment for any cancer
* Use of glucose-lowering agents or a condition that would make a fast from 10:00 pm the evening before until 11:00 am on days 1 and 84 hazardous
* American Urological Association (AUA) total symptom score > 10 or any individual symptom score of greater than or equal to 4
* Psychiatric illness which would prevent compliance with the intervention or would prevent the patient from providing informed consent
* Medical conditions which in the opinion of the treating physician would make this protocol unreasonably hazardous for the participant

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-11; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Clinical toxicity of Se-methyl-seleno-L-cysteine according to the NCI CTCAE version 4.0 | Up to 112 days
  The safety and tolerability data will be summarized using descriptive statistics, by cohort and for all cohorts combined compared to placebo. Reported adverse events will be looked at for possible differences, where appropriate, using graphical methods.
Clinical toxicity of Se-methyl-L-cysteine compared to selenium after multiple doses, according to the NCI CTCAE version 4.0 | Up to 112 days
  The safety and tolerability data will be summarized using descriptive statistics, by cohort and for all cohorts combined compared to placebo. Reported adverse events will be looked at for possible differences, where appropriate, using graphical methods.

SECONDARY OUTCOMES:
Characterization of the pharmacokinetics of Se in the forms Se-methyl-seleno-L-cysteine and selenium at multiple doses | At baseline, and at and .5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 12 hrs after dosing on days 1 and between days 70 and 84
  The pharmacokinetic variables will be tabulated, and descriptive statistics calculated for each cohort, using established pharmacokinetic analysis methods. Plasma and urine pharmacokinetic parameters will be summarized graphically and by arithmetic or geometric means and coefficients of variations for each cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Bergan, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - Roswell Park Cancer Institute, Buffalo, New York
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee